CLINICAL TRIAL: NCT02952274
Title: Comparison Between Ball and Locator Attachments in Patients Receiving Complete Mandibular Overdenture Retained by Single Midline Implant
Brief Title: Ball Vs Locator Attachment in Overdenture Retained by Single Mandibular Implant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Hussein El-Baz, Dr., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1980
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- locater attachment (Active Comparator): mandibular overdenture retained with single midline implant using locator attachment
  Interventions: Device: mandibular overdenture retained with single midline implant using locator attachment
- ball attachment (Active Comparator): mandibular overdenture retained with single midline implant using ball attachment
  Interventions: Device: mandibular overdenture retained with single midline implant using ball attachment

INTERVENTIONS:
Device: mandibular overdenture retained with single midline implant using locator attachment
  Arms: locater attachment
Device: mandibular overdenture retained with single midline implant using ball attachment
  Arms: ball attachment

SUMMARY:
The aim of this study is to compare the ball attachment to the locator attachment regarding the OHRQoL (oral health related quality of life) for completely edentulous patients retaining a mandibular overdenture with a midline placed implant

DETAILED DESCRIPTION:
The selected patients will be informed of the nature of the research work and informed consent will be obtained for each one of them. Only motivated patients who showed co-operation will participate in the study. Patients will be randomly divided into 2 groups.

Conventional upper and lower complete dentures will be constructed before installing the implant where the lower denture will be duplicated into a radiographic stent. CBCT (cone beam computerized tomography) with lower radiographic stent in place stabilized with the upper denture using a rubber base index, will be taken to know the available bone height &width to determine the optimum implant size.

Patients will receive single implant in symphyseal region of mandible. The surgical procedure is carried out under local anaesthesia, following premedication with 2 g amoxicillin (or 600mg of clindamycin) and 1 g paracetamol. After two rinses with 0.2% chlorhexidine gluconate, each lasting 1 min, the labial and lingual mucosa of the anterior mandible is locally infiltrated with 2.2 ml of mepivacaine 2% with 1 : 100,000 adrenalin. The surgical guide made from the duplicated mandibular complete denture is used to mark the implant site.

A crestal incision will be performed and a full-thickness mucoperiosteal flap is raised to expose the anterior mandible. Deep dissection of this flap lingually exposes the cortical plate of the mandible and any lingual concavities. Sequential drilling & implant placement will be the next step. The implant position is adjusted to the midline of the mandible and optimum labiolingual positioning and bone levelling is performed as necessary.

A healing abutment is selected to be 2mm above the mucosa. The mucosa is adjusted and sutured with interrupted sutures (3-0 silk). Postoperatively, the patient should rinse with 0.2% chlorhexidine gluconate mouthwash for 2 weeks. Immediately following implant surgery, generous relief of the existing mandibular complete denture is carried out and a tissue conditioner is applied to the undersurface of the denture. The patient leaves after the surgical operation wearing both the complete maxillary denture opposed by the tissue-conditioned mandibular complete denture. A period of 8 weeks will be allowed for healing and osseointegration.

Then, patients will be recalled for implant loading. The interventional group will receive locator and the control group will receive a standard Ball attachment.

Locator attachment and a ball and socket attachment were randomly assigned to each patient using a computer generated randomization table.

In (Group I) The healing abutment was first removed and the gingival collar irrigated with 0.12% chlorhexidine. The locator attachment was inserted into the implant fixture and torqued to 30 N cm, leaving the attachment base protruding at least 2 mm above the tissue surface. The denture surface of the denture was further relieved to increase the spaces surrounding the attachment assembly and to accommodate the self-curing denture base resin. The denture was inserted after the relief space was filled with resin, and the patient was guided to occlude at centric occlusion. The denture was removed after the resin was cured and adjusted accordingly to assure a comfortable fit.

In (Group2) Patients will receive a standard ball abutment instead of the locator abutment, however the procedures are the same.

Sample Size If there is truly no difference between two groups then 22 patients are required to be 80% sure that the limit of a two sided 90% confidence interval will exclude a difference in means more than 10.

The sample size was done by Sealed Envelope Ltd. 2012

Recruitment

1. Fresh Patient attending in the outpatient clinic in faculty of oral and dental medicine Cairo University will be enrolled in the study
2. Patient from last year records in the outpatient clinic in faculty of oral and dental medicine Cairo University will be contacted by phone and recalled.

Another eligibility examination will be made the researcher and Research will be discussed with all patients and only motivated patient will join the research

1. Sequence generation Is done by computer on the internet by random.org which gives true random numbers
2. Implementation:

Randomized: Computer generated allocation sequence, enrollment and assignment of the participants

Blinding Outcome assessor will be blinded as well as the data analysts for the primary outcome.

It would not be possible to blind the participant or the care provider or the assessor for the second outcome.

Data collection and management:

Data for the primary and secondary outcome will be collected at the day of the surgery and after 3 months on loading of implant and after 6 and 9 months. All data will be saved digitally twice on two separate computers by researcher and the house officer and revised by the supervisor at the end of the data collection.

Participant files are to be stored in numerical order and stored in computer of the removable prosthodontic department

Statistical methods:

Data will be analyzed using IBM (International Business Machines) SPSS advanced statistics (statistical package for social sciences), version 21 (SPSS Inc, Chicago, IL). Numerical data will be described as mean and standard deviation or median and range. Categorical data will be described as numbers and percentages. Data will be explored for normality using kolmogorov-Smirnov test and Shapiro Wilk test. Comparison between two groups for normally distributed numeric variables will be done using the student's t-test while for non normally distributed numeric variables will be done by Mann-Whitney test. Comparisons between categorical variables will be performed using the chi square test. A p-value less than or equal to 0.05 will be considered statistically significant. All tests will be two tailed.

Data Monitoring: data monitoring committee is independent from the sponsor & competing interest. None of the supervisors or the researcher has any conflict of interest with Locator producing companies and is a member of the speaker panel of any company.

Harm: Any complication with implant placement will be reported & managed in the usual way. There is minimal risk of harm associated with the trial.

Auditing: will be independent from the investigator, with every time the data is collected

ELIGIBILITY:
Inclusion Criteria:

1. Completely edentulous patient
2. Patients having enough bone for an implant length of at least 10 mm
3. No apparent bony mal-relation.
4. No intraoral soft and hard tissue pathology
5. No uncontrolled systematic diseases such as hypertension, diabetes and immunodeficiency.

Exclusion Criteria:

1. Drug or alcohol abuse,
2. A health condition precluding surgery,
3. Physical reasons that could affect follow-up,
4. Psychiatric problems,
5. Disorders to the implant area related to a history of radiation therapy to the head and neck, neoplasia, or bone augmentation to the implant site.

Smokers

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
OHRQoL (oral health related quality of life) | 6 months

SECONDARY OUTCOMES:
Peri-implant Plaque index | 6 months
Peri-implant Probing Depth | 6 months

IPD SHARING:
Plan to Share IPD: Yes